CLINICAL TRIAL: NCT06425406
Title: Application of HFNC for the Prevention of Hypoxemia During Perioperative Anesthetic-induced Intubation in Children: A Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HFNC
Record Dates: First submitted 2024-04-15; First posted 2024-05-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: High-flow Nasal Cannula; Children; Pre-oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group HFNC (Experimental): In the HFNC group, the mask ventilation was performed after the patient lost spontaneous breathing until the end-tidal oxygen concentration reached 90 %. The mask was removed and HFNC ( AIRVO2, Fisher Parker Medical Company, Auckland, New Zealand ) was used to record the patient 's safe apnea time. After the end of positive pressure ventilation, intubation or laryngeal mask placement was performed after the end-tidal oxygen concentration reached 90 % or more. During the intubation or placement of the laryngeal mask, the HFNC nasal catheter was kept in the patient 's nose for apnea oxygenation.
  Interventions: Device: high-flow nasal cannula
- Group control (No Intervention): No intervention

INTERVENTIONS:
Device: high-flow nasal cannula — In group H, mask ventilation was performed after the patient lost spontaneous breathing until the end-expiratory oxygen concentration reached 90 %. The lower mask was taken and HFNC was used to record the patient 's safe apnea time.
  Arms: Group HFNC

SUMMARY:
Compared with adults, children have higher metabolic needs, and the airway is more likely to collapse. Before tracheal intubation after anesthesia induction, the patient 's spontaneous breathing completely disappears. At this critical stage, the residual oxygen of the lung is consumed, resulting in hypoxemia and atelectasis. Therefore, it is necessary to explore the best oxygenation strategy during intubation. In addition, ultrasound has become a common equipment in the operating room. It has the advantages of portability, repeatability, and no radiation, and can provide strong support for the diagnosis of gastric distension.

DETAILED DESCRIPTION:
At present, hypoxia is still the main cause of complications and death during perioperative period. Compared with adults, children have lower functional residual volume and lower tolerance to hypoxia caused by apnea due to their special physiological and functional characteristics. During anesthesia induction and tracheal intubation, spontaneous breathing completely disappears. At this critical stage, hypoxemia is prone to occur, which in turn causes various serious complications. Mask ventilation may occur mask ventilation difficulties and flatulence ; since the introduction of nasal high-flow oxygen therapy ( HFNC ) into the operating room in 2015, its oxygenation method has been shown to be able to significantly improve blood oxygen when used alone in pre-oxygenation. When tracheal intubation is performed, HFNC can still maintain ventilation in the patient 's nose, so HFNC can combine the advantages of both masks to perform pre-oxygenation. There are few studies on the effect of HFNC on apnea oxygenation in children in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-10 years old;
* American Society of Anesthesiologists (ASA) Level I or II;
* Children with healthy lungs and hearts;
* Clear headed and able to cooperate with anesthesiologists for treatment.

Exclusion Criteria:

* Contraindications for HFNC: (1) Complete obstruction of the upper respiratory tract; (2) Skull base fracture or nasal bone fracture; (3) Patients who refuse to use HFNC;
* The American Society of Anesthesiologists (ASA) rating is greater than Level II;
* Children with upper respiratory tract infections within 2 weeks;
* Pulmonary dysfunction, congenital heart disease in children;

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Apnoea time | 2-10min
  Investigators will record the time of oxygen saturation drop to 95 % during intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhou, PHD, Study Chair — Henan Provincial People's Hospital
Locations (1):
- Department of Anaesthesiology and Perioperative Medicine, People's Hospital of Zhengzhou University, Henan Provincial People's Hospital, Zhengzhou, Henan, China